CLINICAL TRIAL: NCT04858360
Title: Evaluation of the Effect of Repeated Administration of Topical Local Anaesthetic Mixture of Lidocaine and Prilocaine (EMLA) in a Model of Non-histaminergic Itch Induced by Cowhage.
Brief Title: Inhibition of Non-histaminergic Pruritus Applied Using 3 Different Pruritogens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20200073 1st sub-project
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Drug: Emla 1 hour; Drug: EMLA 3 hours; Other: Vehicle cream for 1 hour; Other: Vehicle cream for 3 hours; Other: Cowhage

INTERVENTIONS:
Drug: Emla 1 hour — At the start of each session, the middle forearms of the subject will each be divided into two squared areas (4x4 cm). On each arm, the two areas will be located 4 cm apart. Then one area will be pre-treated with cutaneous 2.5% lidocaine/2.5% prilocaine cream (EMLA cream) for 1 hour.
Drug: EMLA 3 hours — At the start of each session, the middle forearms of the subject will each be divided into two squared areas (4x4 cm). On each arm, the two areas will be located 4 cm apart. Then one area will be pre-treated with cutaneous 2.5% lidocaine/2.5% prilocaine cream (EMLA cream) for 3 hours.
Other: Vehicle cream for 1 hour — At the start of each session, the middle forearms of the subject will each be divided into two squared areas (4x4 cm). On each arm, the two areas will be located 4 cm apart. Then two area will be pre-treated with a vehicle cream for 1 h.
Other: Vehicle cream for 3 hours — At the start of each session, the middle forearms of the subject will each be divided into two squared areas (4x4 cm). On each arm, the two areas will be located 4 cm apart. Then two area will be pre-treated with a vehicle cream for 3 h.
Other: Cowhage — Cowhage spicules are 1-2 mm in length and have a diameter of 1-3 μm. The spicules are inserted by gently rubbing 30-35 spicules into a 1 cm diameter skin area.

SUMMARY:
With this experiment, we want to use to investigate whether repeated application of EMLA cream as a tool to modulate non-histaminergic itching, which is produced using small needles from the plant mucuna pruriens (it is known that antihistamine does not attenuate this form of itch) and we want to compare the effect of short (1 hour) and prolonged (3 hours) application of EMLA. The sub-project takes place in 3 sessions over a period of 3 consecutive days (24 hours apart). All sessions will be identical.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.).
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamine medications or pain killers.
* Skin diseases
* Hypersensitivity to papaya and mango fruit, cashew nuts and rubber latex
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)
* Known history of anaphylactic shock, or local allergy (contact dermatitis) to lidocaine, prilocaine or other local anaesthetics of the amide type.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Measuring itch intensity by computerized Visual Analog Scale Scoring | For 9 minutes
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable
Measuring pain intensity by computerized Visual Analog Scale Scoring | For 9 minutes
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion measurement | After 1 hour
  Superficial blood perfusion is measured by a Speckle contrast imager
Superficial blood perfusion measurement | After 3 hours
  Superficial blood perfusion is measured by a Speckle contrast imager
Superficial blood perfusion measurement | 10 min after cowhage application
  Superficial blood perfusion is measured by a Speckle contrast imager
Measuring Alloknesis | After 1 hour
  Alloknesis sensation is measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Measuring Alloknesis | After 3 hours
  Alloknesis sensation is measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Measuring Alloknesis | 10 min after cowhage application
  Alloknesis sensation is measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Measuring Hyperknesis | After 1 hour
  Hyperknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Measuring Hyperknesis | After 3 hours
  Hyperknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Measuring Hyperknesis | 10 min after cowhage application
  Hyperknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).

SECONDARY OUTCOMES:
Measuring Erythema | After 1 hour
  The onset of erythema is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Erythema | After 3 hours
  The onset of erythema is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Erythema | 10 min after cowhage application
  The onset of erythema is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Skin Pigmentation | After 1 hour
  The onset of skin pigmentation is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Skin Pigmentation | After 3 hours
  The onset of skin pigmentation is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Skin Pigmentation | 10 min after cowhage application
  The onset of skin pigmentation is measured with a spectrometer (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia lo Vecchio, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark